CLINICAL TRIAL: NCT00257907
Title: Correlation of the Precursor Frequency of CD4 + Effector Memory T Cells With Induration Measured in the Tuberculin Skin Test (TST)
Brief Title: Immune Response to Mycobacterium Tuberculosis Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060030; 06-I-0030
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-02-24

CONDITIONS: Latent Tuberculosis
Keywords: Latent Tuberculosis; PPD; Antigen Specific T-Cells; Lymphocyte Proliferation Assay; HIV; LPA
MeSH Terms: conditions — Latent Tuberculosis

SUMMARY:
This study will examine how the immune system responds to infection with Mycobacterium tuberculosis bacteria (bacteria that cause tuberculosis) in order to better understand how the germ produces infection and how the immune response might work to control the infection.

Only about one in 10 people infected by M. tuberculosis become sick, sometimes years or even decades after exposure. It is not known why some people become sick and most do not, but the immune system of people who never develop disease may be better able to control the bacteria. This study will evaluate the latent form of M. tuberculosis infection to further the understanding of the immune mechanisms - particularly the role of certain white blood cells - involved in the disease process.

Healthy volunteers 18 years of age and older may be eligible for this study. Candidates are screened with a medical history, family history of medical conditions, sexual history, history of drug use, physical examination and blood tests, including a test for HIV. People in Mali, West Africa, and in local health clinics in the United States may participate.

At the start of the study, participants have blood tests and a tuberculin skin test (PPD test), which indicates whether a person has been exposed to tuberculosis bacteria. For the PPD, a tiny amount of liquid containing dead tuberculosis antigen is put under the skin of the forearm with a needle. The antigen cannot cause infection or disease.

After 3 days, participants have another blood test and the site of the tuberculin test is examined for swelling that would indicate a positive result. Participants with a positive PPD have a chest x-ray to check for tuberculosis disease. Those whose x-ray is also positive are withdrawn from the study and referred to their doctor for evaluation and treatment. Those whose x-ray is negative return to the clinic within 3 weeks of the tuberculin test to give another blood sample.

Participants whose PPD is negative have a second tuberculin test 10 to 21 days later and return 3 days after the test to determine if it is still negative or if it is positive. (Some people who are negative after the first test may test positive after the second procedure.) Those whose test is still negative end their participation in the study at that time. Participants whose second PPD is positive have a chest x-ray as described above, and those with a negative chest x-ray return in 3 weeks to donate one last blood sample.

The purpose of the present study is to evaluate the latent form of this infection, the prevalence of which worldwide exceeds that of active disease. Our hypothesis is that in latent tuberculosis antigen specific effector memory CD4+ T cells are responsible for the generation of clinically measurable delayed type hypersensitivity and that central memory CD4+T cells are not directly involved in this process. We base this idea on the assumption that latent tuberculosis is a state of antigen persistence and that effector memory T cells should be maintained as long as antigen/infection is present.

We propose to conduct this study in Mali, West Africa and local clinics in the U.S. Tuberculosis affects 593/100,000(2) individuals in Mali and most have been exposed to the disease. Additionally it would be important to evaluate the same parameters locally as latent infection is one of the major factors for reactivation tuberculosis in this country. Patients would be enrolled in 4 major groups: HIV-/TST- (Group A), HIV-/TST+ (Group B), HIV+/TST+(G roup C) and HIV+/TST- (Group D).

To evaluate this hypothesis we plan to enroll between 100 - 300 patients over the course of 2 years from both countries. Blood samples before and at predetermined time points after the application of Purified Protein Derivative (PPD) will be obtained to determine the fraction of CD4+ T cells which produce interferon gamma in response to stimulation with PPD with a 16hr antigen stimulation assay. Appropriate staining will be done to ascertain the phenotype as well as cytokine production (Interferon gamma,( IFN gamma), Interleukin 2 (IL2) and Tumour Necrosis Factor ( TNF)). Additionally lymphocyte proliferation will be studied using 5-(and-6)-carboxyflouorescein diacetate succinimidyl ester (CFSE.)

In conducting this study we hope to further the understanding of the immune mechanisms involved, particularly mechanisms of T cell memory, which would provide insights into TB and HIV pathogenesis. We also believe that understanding these mechanisms could lead towards establishment of surrogates for immunity in TB vaccine studies, which could enhance vaccine trial design. It might also help in understanding better the immunological dynamics of tuberculosis co-infection in individuals with HIV infection.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a major global health concern. One third of the world's population is infected with Mycobacterium tuberculosis. Two to 3 million people die every year of the disease with 8-10 million new cases per year. It is projected that there will be 90 million new cases and 30 million deaths over the next decade. For a disease, which we know to have existed since 2400 BC, our understanding of its pathogenesis is incomplete, especially in relation to the human immune response and the role of lymphocytes in particular.

The purpose of the present study is to evaluate the latent form of this infection, the prevalence of which worldwide exceeds that of active disease. Our hypothesis is that in latent tuberculosis antigen specific effector memory CD4+ T cells are responsible for the generation of clinically measurable delayed type hypersensitivity and that central memory CD4+T cells are not directly involved in this process. We base this idea on the assumption that latent tuberculosis is a state of antigen persistence and that effector memory T cells should be maintained as long as antigen/infection is present.

We propose to conduct this study in Mali, West Africa and local clinics in the U.S. Tuberculosis affects 593/100,000(2) individuals in Mali and most have been exposed to the disease. Additionally it would be important to evaluate the same parameters locally as latent infection is one of the major factors for reactivation tuberculosis in this country. Patients would be enrolled in 4 major groups: HIV-/TST- (Group A), HIV-/TST+ (Group B), HIV+/TST+ (Group C) and HIV+/TST- (Group D).

To evaluate this hypothesis we plan to enroll between 100 - 300 patients over the course of 2 years from both countries. Blood samples before and at predetermined time points after the application of Purified Protein Derivative (PPD) will be obtained to determine the fraction of CD4+ T cells which produce interferon gamma in response to stimulation with PPD with a 16hr antigen stimulation assay. Appropriate staining will be done to ascertain the phenotype as well as cytokine production (Interferon gamma, ( IFN gamma), Interleukin 2 (IL2) and Tumour Necrosis Factor (TNF)). Additionally lymphocyte proliferation will be studied using 5-(and-6)-carboxyflouorescein diacetate succinimidyl ester (CFSE.)

In conducting this study we hope to further the understanding of the immune mechanisms involved, particularly mechanisms of T cell memory, which would provide insights into TB and HIV pathogenesis. We also believe that understanding these mechanisms could lead towards establishment of surrogates for immunity in TB vaccine studies, which could enhance vaccine trial design. It might also help in understanding better the immunological dynamics of tuberculosis co-infection in individuals with HIV infection.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age18 yrs. or older.
* Adequate venous access.
* Willingness to allow blood samples to be used for future studies of immune function and disease pathogenesis.
* Ability to give informed consent and willingness to comply with study requirements and procedures.
* Willingness to have PPD placed.
* Willingness to undergo HIV testing.

EXCLUSION CRITERIA:

* Hgb less than or equal to 7.9 g/dl
* A known medical disorder or other circumstance which in the opinion of the PI might make the participation of the individual unsafe or difficult.
* Active TB or a history of treated tuberculosis infection.
* Presently suffering from an acute infection.
* History of a severe reaction to PPD application or known allergy to a component of the PPD.
* Severe burns or Eczema.
* PPD less than or equal to 8 weeks previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2005-11-18; Study Completion 2016-02-24

CONTACTS AND LOCATIONS:
Overall Officials: Sophia B Siddiqui, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Mali-NIAID HIV Research Initiative FMPOS, Bamako, Mali

REFERENCES:
- [Background] Kaufmann SH. Protection against tuberculosis: cytokines, T cells, and macrophages. Ann Rheum Dis. 2002 Nov;61 Suppl 2(Suppl 2):ii54-8. doi: 10.1136/ard.61.suppl_2.ii54. PMID 12379623
- [Background] Pais TF, Silva RA, Smedegaard B, Appelberg R, Andersen P. Analysis of T cells recruited during delayed-type hypersensitivity to purified protein derivative (PPD) versus challenge with tuberculosis infection. Immunology. 1998 Sep;95(1):69-75. doi: 10.1046/j.1365-2567.1998.00561.x. PMID 9767459
- [Background] Sallusto F, Geginat J, Lanzavecchia A. Central memory and effector memory T cell subsets: function, generation, and maintenance. Annu Rev Immunol. 2004;22:745-63. doi: 10.1146/annurev.immunol.22.012703.104702. PMID 15032595